CLINICAL TRIAL: NCT04073121
Title: Physician Initiated, Prospective, Non-Randomized Multi-center Trial, Investigating the Safety and Efficacy of the Treatment With Luminor DCB and Angiolite DES of iVascular in TASC C and D Tibial Occlusive Disease in Patients With Critical Limb Ischemia
Brief Title: Investigating the Safety and Efficacy of the Treatment With Luminor DCB and Angiolite DES of iVascular in TASC C and D Tibial Occlusive Disease in Patients With Critical Limb Ischemia
Acronym: MERLION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018/2800
Record Dates: First submitted 2019-08-26; First posted 2019-08-29 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Critical Limb Ischemia
Keywords: Angioplasty; Drug Coated Balloon; Drug Coated Stents
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Luminor DCB and Angiolite DES (Experimental): Study Devices
  Interventions: Device: Luminor DCB and Angiolite DES

INTERVENTIONS:
Device: Luminor DCB and Angiolite DES — Patient to undergo angioplasty with Luminor DCB and Angiolite DES

SUMMARY:
This study aims to evaluate the 12 month outcome of the mono- or combination therapy with iVascular Luminor DCB and Angiolite DES for treatment of TASC C and TASC D long tibial occlusive disease, presenting with critical limb ischemia.

DETAILED DESCRIPTION:
Extensive arterial occlusions significantly reduces distal arterial perfusion, and may eventually lead to Critical Limb Ischemia (CLI). The pathology gives rise to symptoms such as ischemic pain, slow healing wounds at lower extremity and gangrene. It places patients with multi-segment occlusion at high risks of amputations and mortality.

The treatment methods for such long occlusive lesions are limited. Traditionally, the standard of care would be surgical revascularization. This is because lesion length have been identified in several studies as an independent risk factor for the development of restenosis after angioplasty and/or stenting. However, thanks to recent advances in endovascular techniques, such as the utilization of subintimal technique for crossing long segment occlusions, it is now possible to employ endovascular techniques for suitable patients.

The re-establishment of an in-line flow, even if only temporary, can allow tissue healing, which is vital in achieving limb salvage. In addition, the use of Drug Coated Balloons (DCB) and Drug Eluting Stents (DES) can potentially reduce restenosis rate.

To date, there are few studies that have evaluated the performance of DCB in lesions that are longer than 10cm. We hope to evaluate the performance of iVascular Luminor DCB and Angiolite DES when used in the treatment of such lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patient 21 and above
* Patient has critical limb ischemia, presenting a score from 4 to 6 following Rutherford Classification
* Patient is willing to comply with the specified follow-up evaluations at specified time points
* Patient understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
* Patient has a projected life expectancy of at least 12 months
* Prior to enrolment, the guidewire has crossed target lesion
* Patient is eligible for treatment with Luminor Paclitaxel-Eluting Peripheral Balloon Dilation Catheter and Angiolite Drug Eluting Stent
* De novo and post-PTA restenotic lesions located in the tibial arteries suitable for endovascular surgery
* The target lesion is located within the native tibial artery
* The length of the target lesion is >100mm and considered as TASC C or D lesion according to TASC II Classification
* The target lesion has angiographic evidence of stenosis >50% or occlusion, which can be passed with standard guidewire manipulation
* Target vessel diameter visually estimated is >1.5mm and <4.5mm below the knee
* Either one or two different tibial arteries may be treated. Lesions in the treated segment may be continuous or may have gaps present between stenosis and occlusions.
* Any tibial vessel intervened on must have distal reconstitution above the ankle
* Inflow iliac, SFA and popliteal lesions can be treated during the same procedure using standard angioplasty and/or approved device. These inflow lesions must be treated first prior to consideration of the BTK lesion. The patient can be enrolled if the inflow lesions are treated with good angiographic results (must have <30% residual stenosis and no evidence of embolization).
* There is angiographic evidence of at least one-vessel-runoff to the foot, irrespective of whether or not outflow-was established by means of previous endovascular intervention.

Exclusion Criteria:

* Patient refusing treatment
* Patient is permanently wheelchair-bound or bedridden
* Presence of a stent in the target lesions that was placed during a previous procedure
* Untreated flow-limiting inflow lesions
* Any previous surgery in the same limb
* Presence of an aortic thrombosis or significant common femoral ipsilateral stenosis
* Previous bypass surgery in the same limb
* Patient for whom antiplatelet therapy, anticoagulants or thrombolytic drugs are contraindicated.
* Patients who exhibit persistent acute intraluminal thrombus of the proposed lesion site
* Perforation at the angioplasty site evidenced by extravasation of contrast medium
* Patients with known hypersensitivity to heparin, including those patients who have a previous incidence of heparin-induced thrombocytopenia (HIT) type II
* Patients with uncorrected bleeding disorders
* Aneurysm located at the level of SFA/popliteal artery
* Non-atherosclerotic disease resulting in occlusion (e.g. embolism, Buerger's disease, vasculitis)
* Severe medical comorbidities (untreated CFA/CHF, severe COPD, metastatic malignancy, dementia, etc.) or other medical conditions that would preclude compliance with the study protocol or 1-year life expectancy
* Major distal amputation (above the transmetatarsal) in the study limb or non-study limb
* Septicemia or bacteremia
* Patient has undrained pus or spreading wet gangrene in the foot that is not controlled at the time of revascularization procedure.
* Episode of acute limb ischemia within the previous 1 month
* Use of thrombectomy, atherectomy, or laser devices during procedure
* Any patient considered to be hemodynamically unstable at onset of procedure
* Known allergy to contrast media that cannot be adequately pre-medicated prior to the study procedure.
* Patient is participating in another research study of a device, medication, biologic or other agent within 30 days which could in the opinion of the investigator affect the results of this study.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Freedom from Major Adverse Events | 30 days post-operation
  No device- and procedure-related mortality through 30 days, no major target limb amputation.
Freedom from Target Lesion Revascularization | 12 months post-operation
  No re-intervention performed for more than 50% diameter stenosis at the target lesion after documentation of recurrent clinical symptoms of patient.

SECONDARY OUTCOMES:
Primary patency rate | 6 and 12 months post operation
  Absence of hemodynamically significant stenosis on duplex ultrasound (systolic velocity ration no greater than 2.5) at the target lesion and without TLR within the time of procedure and given follow-up
Technical success | immediately post-operation
  Ability to cross and dilate the lesion and achieve residual angiographic stenosis no greater than 30%
Freedom from clinically-driven TLR | 6 month follow-up
  Defined as absence of any repeat intervention to maintain and re-establish patency within the region of the treated arterial vessel plus 5mm proximal and distal to the treated lesion edge
Clinical success at follow-up | 1, 6 and 12 months post-operation
  Improvement of Rutherford Classification

CONTACTS AND LOCATIONS:
Overall Officials: Tjun Yip Tang, Principal Investigator — Singapore General Hospital
Locations (2):
- Singapore (2):
  - Singapore General Hospital, Singapore
  - Khoo Teck Puat Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baril DT, Marone LK, Kim J, Go MR, Chaer RA, Rhee RY. Outcomes of endovascular interventions for TASC II B and C femoropopliteal lesions. J Vasc Surg. 2008 Sep;48(3):627-33. doi: 10.1016/j.jvs.2008.04.059. PMID 18727966
- [Background] Christenson BM, Rochon P, Gipson M, Gupta R, Smith MT. Treatment of infrapopliteal arterial occlusive disease in critical limb ischemia. Semin Intervent Radiol. 2014 Dec;31(4):370-4. doi: 10.1055/s-0034-1393974. No abstract available. PMID 25435663
- [Background] Giles KA, Pomposelli FB, Spence TL, Hamdan AD, Blattman SB, Panossian H, Schermerhorn ML. Infrapopliteal angioplasty for critical limb ischemia: relation of TransAtlantic InterSociety Consensus class to outcome in 176 limbs. J Vasc Surg. 2008 Jul;48(1):128-36. doi: 10.1016/j.jvs.2008.02.027. Epub 2008 May 23. PMID 18502084
- [Background] TASC Steering Committee; Jaff MR, White CJ, Hiatt WR, Fowkes GR, Dormandy J, Razavi M, Reekers J, Norgren L. An Update on Methods for Revascularization and Expansion of the TASC Lesion Classification to Include Below-the-Knee Arteries: A Supplement to the Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). Vasc Med. 2015 Oct;20(5):465-78. doi: 10.1177/1358863X15597877. Epub 2015 Aug 12. PMID 26268268
- [Background] Soderstrom MI, Arvela EM, Korhonen M, Halmesmaki KH, Alback AN, Biancari F, Lepantalo MJ, Venermo MA. Infrapopliteal percutaneous transluminal angioplasty versus bypass surgery as first-line strategies in critical leg ischemia: a propensity score analysis. Ann Surg. 2010 Nov;252(5):765-73. doi: 10.1097/SLA.0b013e3181fc3c73. PMID 21037432
- [Background] Clark TW, Groffsky JL, Soulen MC. Predictors of long-term patency after femoropopliteal angioplasty: results from the STAR registry. J Vasc Interv Radiol. 2001 Aug;12(8):923-33. doi: 10.1016/s1051-0443(07)61570-x. PMID 11487672
- [Background] Zeller T, Rastan A, Macharzina R, Tepe G, Kaspar M, Chavarria J, Beschorner U, Schwarzwalder U, Schwarz T, Noory E. Drug-coated balloons vs. drug-eluting stents for treatment of long femoropopliteal lesions. J Endovasc Ther. 2014 Jun;21(3):359-68. doi: 10.1583/13-4630MR.1. PMID 24915582